CLINICAL TRIAL: NCT04029116
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Oral Ibrexafungerp (SCY-078) Compared to Placebo in Subjects With Recurrent Vulvovaginal Candidiasis (VVC)
Brief Title: Phase 3 Study of Oral Ibrexafungerp (SCY-078) Vs. Placebo in Subjects With Recurrent Vulvovaginal Candidiasis (VVC)
Acronym: CANDLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SCY-078-304
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Vulvovaginal Candidiasis
Keywords: Recurrent yeast infection; Recurrent yeast vaginitis; Chronic yeast vaginitis; Ibrexafungerp; SCY-078; RVVC
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Fluconazole; ibrexafungerp

STUDY DESIGN:
Intervention Model Description: Open label (acute phase treatment) followed by Randomized, Double Blinded phase
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibrexafungerp (Experimental): Oral Fluconazole 150 mg every 72 hours for 3 doses followed by Oral Ibrexafungerp 300 mg BID (one day) every 4 weeks for a total of 6 dosing days
  Interventions: Drug: Fluconazole Tablet; Drug: IBREXAFUNGERP
- Placebo (Placebo Comparator): Oral Fluconazole 150 mg every 72 hours for 3 doses followed by Oral Placebo BID (one day) every 4 weeks for a total of 6 dosing days
  Interventions: Drug: Fluconazole Tablet; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Fluconazole Tablet — 150 mg every 72 hours for 3 doses
Drug: IBREXAFUNGERP — 300 mg BID (one day) every 4 weeks for a total of 6 dosing days
  Other Names: SCY-078
  Arms: Ibrexafungerp
Drug: Placebo oral tablet — BID (one day) every 4 weeks for a total of 6 dosing days
  Arms: Placebo

SUMMARY:
This study is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of oral ibrexafungerp (formerly "SCY-078") compared to placebo in female subjects 12 years and older with recurrent VVC (RVVC).

DETAILED DESCRIPTION:
This study is a Phase 3, multicenter, randomized, double-blind study to evaluate the efficacy and safety of oral ibrexafungerp (formerly "SCY-078") compared to placebo in female subjects 12 years and older with RVVC. The primary objective of the study is to evaluate the efficacy of oral ibrexafungerp in preventing recurrences of VVC in subjects with RVVC based on Clinical Success. Approximately 320 subjects are planned to be enrolled into the study. All subjects will receive treatment with oral fluconazole for their acute episode present at screening. Subjects who respond to fluconazole for their acute episode will be enrolled in the prevention of recurrence phase of the study and randomized to ibrexafungerp or placebo.

Subjects who fail treatment with fluconazole for their acute episode will be included in a nested open label Sub-Study, in which they will be offered one-day oral ibrexafungerp for their unresolved acute episode.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of symptomatic VVC with microscopic examination with KOH positive for yeast and normal vaginal pH.
* History of 3 or more episodes of VVC in the past 12 months.
* Culture confirmation and resolution of the signs and symptoms of the initial VVC episode (with treatment).
* Able to take oral tablets and capsules.

Key exclusion Criteria:

* Vaginal conditions other than recurrent VVC that may interfere with the diagnosis or evaluation of response to therapy.
* Recent use of systemic and/or topical vaginal antifungal products.
* Pregnant.
* History of major system organ disease.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 440 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nkechi Azie, MD, Study Director — Scynexis, Inc.
Locations (25):
- United States (25):
  - Precision Trials LLC, Phoenix, Arizona
  - Women's Healthcare Research Corp, San Diego, California
  - Altus Research - Hunt - PPDS, Lake Worth, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Healthcare Clinical Data Inc, North Miami, Florida
  - Clinical Research Prime - ClinEdge - PPDS, Idaho Falls, Idaho
  - Clinical Trials Management, Covington, Louisiana
  - Women Under Study, LLC, New Orleans, Louisiana
  - Unified Women's Clinical Research, Hagerstown, Maryland
  - Wayne State University, Detroit, Michigan
  - Center For Women's Health and Wellness LLC, Lawrenceville, New Jersey
  - Lawrence Obstetrics Gynecology Clinical Research LLC, Lawrenceville, New Jersey
  - Bosque Women's Care, Albuquerque, New Mexico
  - Carolina Women's Research and Wellness Center, Durham, North Carolina
  - Unified Womens CLinical Research, Greensboro, North Carolina
  - Unified Women's Clinical Research Raleigh, Raleigh, North Carolina
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - Group For Women, Winston-Salem, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Obstetrics and Gynecology Associates of Erie, PC, Erie, Pennsylvania
  - Jefferson University Hospital, Philadelphia, Pennsylvania
  - Chattanooga Medical Research Inc, Chattanooga, Tennessee
  - Medical Research Center of Memphis, LLC, Memphis, Tennessee
  - TMC Life Research Inc, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 49 medical centers between 21Oct2019 and 29Nov2021
Pre-assignment Details: 440 subjects were enrolled into the acute phase of the study with 156 of them discontinuing. 260 then entered into the recurrence phase
Period: Overall Study
Arm/Group | Ibrexafungerp | Placebo
Started | 130 | 130
Discontinued | 12 | 16
Completed | 118 | 114
Not Completed | 12 | 16
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 3 | 5
Not completed — Physician Decision | 2 | 0
Not completed — Pregnancy | 1 | 2
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibrexafungerp | Placebo | Total
Number analyzed (Participants) | 130 | 130 | 260
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 129 | 130 | 259
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (10.23) | 33.7 (9.29) | 33.9 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 130 | 260
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 10 | 22
  Not Hispanic or Latino | 118 | 120 | 238
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 12 | 21
  White | 120 | 114 | 234
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 43 | 85
  Bulgaria | 37 | 35 | 72
  Poland | 17 | 14 | 31
  Russia | 34 | 38 | 72

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success
Description: Efficacy as measured by the percentage of subjects with documented Clinical Success.
Time Frame: Week 24
Population: Intent-to-Treat Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp | Placebo
Number analyzed (Participants) | 130 | 130
Participants
  Clinical Success | 85 | 69
  Clinical Failure | 45 | 61

2. Secondary Outcome: The Percentage of Subjects With no Mycologically Proven Recurrence
Description: Efficacy as measured by the percentage of subjects with no Mycologically Proven Recurrence
Time Frame: Week 24
Population: Intent-to-Treat Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp | Placebo
Number analyzed (Participants) | 130 | 130
Participants
  No Mycologically Proven Recurrence | 92 | 76
  Mycologically Proven Recurrence | 38 | 54

3. Secondary Outcome: Safety and Tolerability
Description: Safety as measured by the number of subjects who discontinue due to treatment related adverse events.
Time Frame: Week 24
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp | Placebo
Number analyzed (Participants) | 130 | 130
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: up to 38 weeks
Arm/Group | Ibrexafungerp | Placebo
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/130
Serious Adverse Events (participants affected / at risk) | 1/130 | 0/130
Other Adverse Events (participants affected / at risk) | 66/130 | 41/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrexafungerp (N=130) | Placebo (N=130)
COVID-19 (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrexafungerp (N=130) | Placebo (N=130)
Diarrhoea (Gastrointestinal disorders) | 10 | 5
Nausea (Gastrointestinal disorders) | 7 | 5
Abdominal pain upper (Gastrointestinal disorders) | 7 | 4
Bacterial vaginosis (Infections and infestations) | 10 | 11
COVID-19 (Infections and infestations) | 7 | 5
Headache (Nervous system disorders) | 25 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT04029116/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT04029116/SAP_001.pdf